CLINICAL TRIAL: NCT00880646
Title: Effects of the Combination of L-Arabinose and Indigestible Dextrin on Obesity: a Double-Blind, Randomized Controlled Trial
Brief Title: Effects of the Combination of L-Arabinose and Indigestible Dextrin on Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: Unitika Ltd. (Industry)
Responsible Party: Fumiko Higashikawa, PhD/Associate professor, Hiroshima University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: eki-124
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: Oolong tea containing L-arabinose and indigestible dextrin
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Oolong tea (Placebo)

INTERVENTIONS:
Dietary Supplement: Oolong tea containing L-arabinose and indigestible dextrin
  Arms: 1
Dietary Supplement: Oolong tea (Placebo)
  Arms: 2

SUMMARY:
This study aims to investigate the effect of supplement containing L-arabinose and indigestible dextrin on body mass index, body fat mass, abdominal circumference, visceral fat mass, and serum biochemical parameters in overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as based on medical history and physical examination
* BMI between 25 and 30 kg/m2
* Willing not to serve as blood donor during the study
* Informed consent signed

Exclusion Criteria:

* Female subjects who are pregnant or nursing a child
* Participation in any clinical trial up to 90 days before Day 01 of this study
* Renal or hepatic dysfunction
* Heart disease
* Under medication
* Subjects who are taking functional food designed for weight loss or serum lipid reduction

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-03; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Body mass index | 20 weeks

SECONDARY OUTCOMES:
Body fat mass | Every 4 weeks (Overall 20 weeks)
Abdominal circumference | Every 4 weeks (Overall 20 weeks)
Visceral fat area by CT scan | Week 0, Week 12
Serum lipid profile | Every 4 weeks (Overall 20 weeks)
Serum adiponectin and leptin levels | Week 0, Week 12
Fasting serum glucose and HbA1c levels | Every 4 weeks (Overall 20 weeks)
Frequency of bowel movement | 20 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hiroshima University, Hiroshima, Hiroshima, Japan